CLINICAL TRIAL: NCT03329274
Title: Registry for Patients With Erdheim-Chester Disease and Other Histiocytoses
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17-516
Record Dates: First submitted 2017-10-26; First posted 2017-11-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Erdheim-Chester Disease
Keywords: registry; Other Histiocytoses; Langerhans cell histiocytosis; Rosai Dorfman disease; 17-516
MeSH Terms: conditions — Erdheim-Chester Disease; Histiocytosis, Langerhans-Cell; Histiocytosis, Sinus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Erdheim-Chester Disease and Other Histiocytoses

SUMMARY:
The investigators want to understand more about what kinds of health problems are caused by histiocytosis, what happens as a result of different treatments, and how ECD affects people's lives, their feelings and their attitudes. The investigators also want to learn how these things change over time for people with these conditions. To try to figure this out, doctors would like to collect information about people who have histiocytosis and how they are treated for this disease.

Some participants will be asked to complete a brief interview over the telephone. Only a limited number of interviews will take place, and not everyone will be asked to participate in the interview. It is okay if the participant does not want to participate in the interview portion. If this is the case, the participant should let the study team member know when contacted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Erdheim-Chester Disease, Langerhans cell histiocytosis, Rosai Dorfman disease, or another histiocytic neoplasm by either 1) documented histopathologic establishing ECD or HN or 2) documented histopathologic findings compatible with Erdheim-Chester disease or HN in the context of corroborating clinical and/or radiologic findings or 3) documented radiologic findings, in the absence of a biopsy having been performed or yielding evaluable tissue, that are felt by the Principal Investigator to unequivocally represent an ECD/HN diagnosis given the clinical context or 4) self reported with supporting documentation upon medical record collection.
* Proficiency in English, in the determination of the Investigator or by self report.
* Willing to have historical and future HN-related health records sent to Registry review.

Exclusion Criteria:

* Patients unwilling to sign consent.
* Participants under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Erdheim-Chester Disease and other HN will be enrolled in this registry study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-10-26 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Create registry for Erdheim-Chester Disease and Other Histiocytoses | 3 years
  This ECD and Other Histiocytoses registry is motivated to capture comprehensive clinical information as well as patient-centered data about ECD and Other Histiocytoses patients.

CONTACTS AND LOCATIONS:
Overall Officials: Eli Diamond, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Reiner AS, Alici Y, Correa DD, Bossert D, Sigler AM, Fournier D, Brewer K, Goyal G, Atkinson TM, Marathe P, Mao JJ, Panageas KS, Diamond EL. Anxiety and depression in patients with histiocytic neoplasms and their associated clinical features. Blood Adv. 2025 Mar 25;9(6):1376-1386. doi: 10.1182/bloodadvances.2024014850. PMID 39626273
- [Derived] Kirchner J, Hatzoglou V, Buthorn JB, Bossert D, Sigler AM, Reiner AS, Ulaner GA, Diamond EL. 18F-FDG PET/CT versus anatomic imaging for evaluating disease extent and clinical trial eligibility in Erdheim-Chester disease: results from 50 patients in a registry study. Eur J Nucl Med Mol Imaging. 2021 Apr;48(4):1154-1165. doi: 10.1007/s00259-020-05047-8. Epub 2020 Oct 15. PMID 33057928
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm